CLINICAL TRIAL: NCT00003116
Title: Allogeneic Peripheral Blood Progenitor Cell Transplantation Using Histocompatible Sibling-Matched Donor Cells After High-Dose Busulfan/Cyclophosphamide as Therapy for Hematologic Malignancies
Brief Title: High-Dose Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hillard Lazarus, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1995T; P30CA043703 (NIH); CASE-CWRU-1995; NCI-G97-1354; CASE1995T (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; recurrent/refractory childhood Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cyclosporine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — Filgrastim (G-CSF) is administered subcutaneously twice a day beginning 3 hours after completion of cell infusion and continuing until blood counts recover.
Drug: busulfan — high-dose oral busulfan every 6 hours on days -8 to -5
Drug: cyclophosphamide — cyclophosphamide IV twice a day on days -4 and -3
Drug: cyclosporine — cyclosporine IV over 6 hours on day -1 and then 10 hours on day 0 for 2 doses (allogeneic only)
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation — Allogeneic peripheral blood progenitor cells IV are administered on day 0.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving busulfan, cyclophosphamide, and filgrastim together with peripheral stem cell transplantation from a sibling donor works in treating patients with hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of using allogeneic peripheral blood progenitor cell infusions obtained from normal histocompatible sibling donors for reconstituting bone marrow and immunologic function when given after high-dose busulfan/cyclophosphamide in patients with a hematologic malignancy.
* Determine the efficacy of this treatment in these patients.
* Determine the ability to mobilize hematopoietic progenitor cells from normal donors given filgrastim (G-CSF) by determining the hematopoietic progenitor cell content of allogeneic peripheral blood progenitor cell collections.
* Determine the incidence of engraftment failures in these patients.
* Determine the incidence of severe acute graft-versus-host disease in these patients.

OUTLINE: Patients receive high-dose oral busulfan every 6 hours on days -8 to -5, cyclophosphamide IV twice a day on days -4 and -3, and cyclosporine IV over 6 hours on day -1 and then 10 hours on day 0 for 2 doses (allogeneic only). Allogeneic peripheral blood progenitor cells IV are administered on day 0.

Filgrastim (G-CSF) is administered subcutaneously twice a day beginning 3 hours after completion of cell infusion and continuing until blood counts recover.

Patients are followed every month for 2 months, every 3 months for 6 months, and then every 6 months until disease progression.

PROJECTED ACCRUAL: A total of 40 patients will be accrued over a 15 month period.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically diagnosed:

  * Acute myeloid leukemia in first, second, or third complete remission or first or second early relapse
  * Acute lymphoblastic leukemia in first, second, or third complete remission or first or second early relapse
  * Hodgkin's lymphoma in second or third remission or first, second, or third relapse, or refractory
  * Non-Hodgkin's lymphoma in second or third remission or first, second, or third relapse, or refractory
  * Multiple myeloma and plasma cell leukemia in second or third remission or first, second, or third relapse, or refractory
  * Myelodysplastic syndrome deemed suitable for allogeneic bone marrow transplantation
* No symptoms or signs of CNS involvement and CNS is disease free on lumbar puncture and brain CT scan
* No active meningeal cancer

PATIENT CHARACTERISTICS:

Age:

* 4 to 55 (4 to 60 if donor is identical twin)

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* SGOT/SGPT less than 3 times normal
* Bilirubin less than 2.0 mg/dL

Renal:

* Creatinine less than 2.1 mg/dL
* Creatinine clearance at least 60 mL/min (no greater than 1.5 times normal for children under 40 kg)

Cardiovascular:

* No uncontrolled hypertension
* No uncontrolled congestive heart failure
* No active angina pectoris requiring nitrates
* At least 6 months since prior myocardial infarction
* No major ventricular arrhythmia
* Left ventricular ejection fraction at least 45% on MUGA

Pulmonary:

* No severe or symptomatic restrictive or obstructive lung disease
* FEV_1 greater than 50% of predicted
* DLCO greater than 50% of predicted

Neurologic:

* No severe central or peripheral neurologic abnormality

Other:

* Must have HLA-A,B,C,D/DR identical sibling age 4 to 65, in good health
* No insulin-dependent diabetes mellitus
* No major thyroid or major adrenal dysfunction
* No active infection
* No other active malignancy
* Not pregnant
* HIV negative
* HTLV-I and HTLV-II negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No excessive anthracycline exposure, unless endomyocardial biopsy shows less than grade 2 drug effect and cardiac scan shows at least 50% ejection fraction
* At least 1 year since prior autologous bone marrow or peripheral blood progenitor cell transplant or allogeneic bone marrow transplant

Chemotherapy:

* At least 3 weeks since prior chemotherapy
* No prior excessive carmustine and bleomycin

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent nitroglycerin for angina pectoris
* No concurrent anti-arrhythmic drugs for major ventricular dysrhythmias

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 1997-05; Primary Completion 2006-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Hematopoietic reconstitution measured daily during transplant | at months 2, 4, 7, and 10, and then every 6 months until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Hillard M. Lazarus, MD, Study Chair — Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hosptials Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States